CLINICAL TRIAL: NCT05313425
Title: Effect of Ectoine on Stromal Haze, Wound Healing and Pain After Photorefractive Keratectomy.
Brief Title: Effect of Ectoine After Photorefractive Keratectomy (PRK).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Elkadim, Lecturer of ophthalmology, Tanta University
Other Study IDs: Ectoine after PRK
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Photorefractive Keratectomy; Corneal Haze
Keywords: PRK, surface ablation, corneal haze
MeSH Terms: conditions — Corneal Opacity | interventions — Ophthalmic Solutions; ectoine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ectoine Eye: The right eye of the studied group will be given 2% Ectoine containig , 0.2% sodium hyaluronate eye drops(Ectohylo) hourly.
  Interventions: Other: Ectohylo (R) eye drops
- Control eye: The left eye of the studied group will be give Carboxymethyl cellulose, 0.2% sodium hyaluronate eye drops(Polyfresh Extra) hourly.

INTERVENTIONS:
Other: Ectohylo (R) eye drops — using Ectohylo eye drops post operative after PRK in the right eyes of the patients
  Other Names: Ectoine 2% eye drops
  Groups: Ectoine Eye

SUMMARY:
This is a comparative, open label, parallel group, non interventional study aims to assess the effect of Ectoine containing eye drops on stromal haze, pain and epithelial healing after Photorefractive keratectomy (PRK). The patient apply Ectohylo eye drops (Ectoine +Sodium Hyauronate) in the right eye and Polyfresh Extra eye drops (Carboxymethyl cellulose + Sodium Hyauronate ) in the left eye plus the routine post PRK treatment in both eyes. Post operative pain , epithelial healing and corneal densitometry is observed in both eyes.

DETAILED DESCRIPTION:
Photorefractive keratectomy (PRK) is a commonly used operation for laser vision correction. The main fears of this type of laser vision correction is corneal haze, delayed epithelial healing and postoperative severe pain. Ectoine is a natural compound that has the ability to protect biological membranes from damage and environmental effects. This study assess the use of Ectoine containing eye drops to protect the bare ocular surface and reduce inflammation after PRK that will inturn is expected to affect the post operative corneal haze, pain, and epithelial healing .

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing PRK for myopia and myopic astigmatism when astigmatism is 2.5 diopters or less and myopia with spherical equivalent -4 or less.

Exclusion Criteria:

* patient spherical equivalent more myopic than -4 diopters
* Patients with astigmatism more than 2.5 diopter
* Patients with anisometropia ( difference > 2 diopters)
* Patient with previous ocular surgery
* Patients with chronic systemic disease that can affect results of laser vision correction (e.g. rheumatoid arthritis)
* Pregnant and lactating females

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient enrolled for photorefractive keratectomy for correction of myopia and myopic astigmatism.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Corneal Densitometry (assesed by Pentacam). | 3 months post operative
  Post photo refractive keratectomy early haze (3 months after operation) assesed by Pentacam densitometry

SECONDARY OUTCOMES:
Pain score (0 -10) | 2 days
  pain in the first 2 days post operative (graded 0 to 10)
Time of Epithelial healing (days) | 2-7 days
  Time required for epithelial healing after PRK in days

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elkadim, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in Cornea. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication for 5 months
Access Criteria: Authorized Ophthalmologists specialized in cornea and refractive surgery